CLINICAL TRIAL: NCT01070316
Title: Everolimus (RAD001) Therapy for Epilepsy in Patients With Tuberous Sclerosis Complex
Brief Title: Everolimus (RAD001) Therapy for Epilepsy in Patients With Tuberous Sclerosis Complex (TSC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0998
Record Dates: First submitted 2010-02-15; First posted 2010-02-18 (Estimated); Results first posted 2016-09-23 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-02

CONDITIONS: Epilepsy; Tuberous Sclerosis Complex
Keywords: Epilepsy; Tuberous Sclerosis Complex; Everolimus; RAD001; Mammalian Target of Rapamycin (MTOR)
MeSH Terms: conditions — Epilepsy; Tuberous Sclerosis; Hereditary Sensory and Autonomic Neuropathies | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): Subjects will be administered study drug if they meet study criteria after 4 weeks of baseline phase. The starting dose will be 5 mg/m2/day, rounded to the nearest 2.5 mg/dose, to be taken daily.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus is available in tablet form. The starting dose will be 5 mg/m2/day, rounded to the nearest 2.5 mg/dose, to be taken daily. After two weeks, serum trough level will be measured and dose adjusted according to the following algorithm If Blood trough level is less than 2.5 ng/ml than increase dose by 5 mg/m2/day; If Blood trough level is 2.5-5.0 ng/ml than increase dose by 2.5 mg/m2/day; If Blood trough level is 5.1-10.0 ng/ml than increase dose by 0 mg/m2/day (no change); If Blood trough level is 10.1-15.0 ng/ml than decrease dose by 2.5 mg/m2/day
  Other Names: RAD001; Certican; Afinitor

SUMMARY:
The goal of this study is to learn if the study drug RAD001 can reduced the number of epileptic seizures, and can be taken safety by people who have epilepsy associated with Tuberous Sclerosis Complex.

DETAILED DESCRIPTION:
Tuberous sclerosis complex (TSC) is a genetic disorder with an incidence at birth of 1 in 6000. This disorder is characterized by the development of benign tumors in multiple organ systems, including the brain. The primary neurological manifestations of TSC are epilepsy, mental retardation and autism. Epilepsy is most common, occurring in 80-90% of patients, and often the seizures are severe, unremitting, and uncontrolled by current anticonvulsant medications. It is generally accepted that the seizures arise from cortical and subcortical tubers and surrounding tissue in the brain. These tubers are caused by mutations in the tumor suppressor genes TSC1 or TSC2. The protein products of these genes, hamartin and tuberin, act as negative regulators of the PI3K/PKB(Akt)/mTOR signaling pathway that regulates cell growth and proliferation Everolimus is an immunosuppressant drug that also inhibits mTOR signaling and is capable of reversing aberrant mTOR-dependent effects that occur when hamartin or tuberin are absent or defective. Thus, we hypothesize that drugs like everolimus may be therapeutically useful for the treatment of refractory epilepsy in patients with TSC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals aged two years and older.
* History of epilepsy and at least eight reported seizures in previous 30 days prior to informed consent
* Failure of two or more approved antiepileptic drug therapies
* Clinically definite diagnosis of tuberous sclerosis (modified Gomez criteria or positive genetic test)
* Parents/Caregivers are English-speaking (primary or secondary language acceptable)
* If female and of child bearing potential, documentation of negative pregnancy test at time of informed consent. Sexually active pre-menopausal female or male patients must use adequate contraceptive measures, excluding use of estrogen-containing birth control contraceptive regimen while on study medication. Prior hysterectomy, tubal ligation, complete abstinence, barrier methods which include both a cervical diaphragm and spermicidal jelly, intrauterine devices (IUD), progesterone based contraceptives, or vasectomy in partner are all acceptable forms of contraception
* Adequate bone marrow function as shown by ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, and Hb >9 g/dL
* Adequate liver function as shown by serum bilirubin ≤ 1.5 x upper limit of normal (ULN), ALT and AST ≤ 2.5x ULN, INR and PTT ≤1.5. (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for >2 weeks at time of randomization.)
* Adequate renal function as shown by a serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication

Exclusion Criteria:

* Significant hematological or hepatic abnormality (i.e., transaminase levels > 2.5 x ULN or serum bilirubin >1.5 x ULN, Hemoglobin < 9 g/dL, platelets < < 100 X 109/L , absolute neutrophil count < 1.5 x 109/L)
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks prior to informed consent
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed
* Patients should not receive immunization with attenuated live vaccines within one week of informed consent or during study period
* Patients with coexisting malignancies within past 3 years, except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York heart Association Class III or IV, unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * Severely impaired lung function defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air and/or requirement for continuous supplemental O2
  * Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
  * Active (acute or chronic) or uncontrolled severe infections
  * Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis

    * A known history of HIV seropositivity
    * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
    * Patients with an active, bleeding diathesis
    * Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.
    * Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
    * Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycin (sirolimus, temsirolimus) or to its excipients
    * History of noncompliance to medical regimens

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Krueger, M.D. Ph.D, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Krueger DA, Wilfong AA, Holland-Bouley K, Anderson AE, Agricola K, Tudor C, Mays M, Lopez CM, Kim MO, Franz DN. Everolimus treatment of refractory epilepsy in tuberous sclerosis complex. Ann Neurol. 2013 Nov;74(5):679-87. doi: 10.1002/ana.23960. Epub 2013 Sep 10. PMID 23798472

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 participants were screened; 3 participants were not eligible to begin treatment and were not enrolled
Period: Main Phase
Arm/Group | Everolimus
Started | 20
Completed | 20
Not Completed | 0
Period: Extension Phase
Arm/Group | Everolimus
Started | 18 (Two participants did not qualify for Extension Phase as defined by protocol)
Completed | 14
Not Completed | 4
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 20 study subjects were consented, screened, enrolled, and received study drug
Groups:
- Everolimus: Main Study Phase:
  Subjects will be administered study drug if they meet study criteria after 4 weeks of baseline phase. The starting dose will be 5 mg/m2/day, rounded to the nearest 2.5 mg/dose, taken daily.
  Everolimus: Everolimus is available in tablet form. The starting dose will be 5 mg/m2/day, rounded to the nearest 2.5 mg/dose, to be taken daily. After two weeks, serum trough level will be measured and dose adjusted according to the following algorithm If trough level is less than 2.5 ng/ml than increase dose by 5 mg/m2/day; If trough level is 2.5-5.0 ng/ml than increase dose by 2.5 mg/m2/day; If trough level is 5.1-10.0 ng/ml than increase dose by 0 mg/m2/day (no change); If trough level is 10.1-15.0 ng/ml than decrease dose by 2.5 mg/m2/day
  Following the 4 week titration, subjects will continue in an 8 week maintenance period.
  If subjects qualify for the Extension Phase of the study, they will continue on study drug and be followed through 48 months.
Arm/Group | Everolimus
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Seizure Frequency
Description: The primary efficacy endpoint was the percentage of participants demonstrating a 50% or greater reduction in seizure frequency at the end of the maintenance phase (weeks 13-16) compared to baseline (weeks 1-4)
Time Frame: Baseline (Weeks 1-4), Week 16
Measure: Number; unit: percentage
Arm/Group | Everolimus
Number analyzed (Participants) | 20
percentage | 60

2. Primary Outcome: Number of Participants Continuing Study Medication Over Time
Time Frame: Individual subjects will be assessed every 6 months for up to 48 months; aggregate analysis will take place at end of study
Measure: Number; unit: participants
Arm/Group | Everolimus
Number analyzed (Participants) | 20
participants
  16 weeks | 20
  Entered Extension Phase (4 months) | 18
  6 months | 18
  12 months | 17
  18 months | 16
  24 months | 16
  30 months | 16
  36 months | 15
  42 months | 14
  48 months | 14

ADVERSE EVENTS:
Time Frame: 5 years and 4 months
Arm/Group | Everolimus
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=20)
Infection - URI/Sinus/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Infection - GU (Renal and urinary disorders) | 1 (1)
Infection - GI (Gastrointestinal disorders) | 1 (1)
Infection - unspecified (Infections and infestations) | 1 (1)
Infection - Otitis (Ear and labyrinth disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=20)
Abrasion (Skin and subcutaneous tissue disorders) | 4 (5)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
ADHD (Psychiatric disorders) | 1 (1)
Agitation/Irritability (Psychiatric disorders) | 8 (12)
Allergic Rhinitis (General disorders) | 1 (1)
Allergic conjunctivitis (Eye disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 3 (6)
Ataxia (Nervous system disorders) | 1 (1)
Back pain (General disorders) | 1 (1)
Bruising (General disorders) | 2 (2)
Cheilitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cholesterol (Investigations) | 3 (4)
Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 4 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 8 (23)
Ear Pain (Ear and labyrinth disorders) | 2 (2)
Edema (Blood and lymphatic system disorders) | 2 (5)
Fatigue (General disorders) | 4 (7)
Fever (General disorders) | 9 (18)
Flu-like symptoms (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 5 (9)
Gastrointestinal Other (Gastrointestinal disorders) | 2 (2)
Headache (General disorders) | 5 (5)
Hemorrhage (Blood and lymphatic system disorders) | 3 (3)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperkalemia (Investigations) | 1 (1)
Hypoalbuminemia (Investigations) | 1 (1)
Hypokalemia (Investigations) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Hypophosphatemia (Investigations) | 1 (1)
Infection - Conjunctivitis (Eye disorders) | 2 (2)
Infection - GI (Gastrointestinal disorders) | 10 (22)
Infection - GU (Renal and urinary disorders) | 4 (6)
Infection - Lymphatics (Blood and lymphatic system disorders) | 1 (1)
Infection - Otitis (Ear and labyrinth disorders) | 11 (26)
Infection - Skin (Skin and subcutaneous tissue disorders) | 9 (21)
Infection - Unspecified (Infections and infestations) | 3 (3)
Infection - URI/Sinus/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 20 (131)
Insomnia (General disorders) | 6 (9)
Laboratory - Other (Investigations) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 4 (6)
Leg pain (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Metabolic - Other (Investigations) | 1 (1)
Mucositis/Atomatitis (Gastrointestinal disorders) | 17 (78)
Muscle pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal - other (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophils - other (Blood and lymphatic system disorders) | 4 (16)
Osteopenia/Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Other (Immune system disorders) | 1 (1)
Other (Skin and subcutaneous tissue disorders) | 5 (5)
Otitis media (Ear and labyrinth disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 9 (12)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sialorrhea (Gastrointestinal disorders) | 1 (2)
Somnolence (General disorders) | 1 (1)
Speech impairment (General disorders) | 2 (2)
Sprain/Strain/Soft tissue (Musculoskeletal and connective tissue disorders) | 5 (6)
Stye (Eye disorders) | 1 (1)
Teeth (Gastrointestinal disorders) | 2 (2)
Thirst (Gastrointestinal disorders) | 2 (2)
Throat pain (Gastrointestinal disorders) | 1 (1)
Transaminase (Investigations) | 2 (9)
Unspecified pain (General disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal itching (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (22)
Weight loss (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No